CLINICAL TRIAL: NCT04744077
Title: Physical Activity and Social-media Support
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State Polytechnic University, Pomona (Other)
Responsible Party: Principal Investigator, Zakkoyya Lewis-Trammell, Assistant Professor, California State Polytechnic University, Pomona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-21-8
Record Dates: First submitted 2021-01-29; First posted 2021-02-08 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Trust
Keywords: social media; physical activity; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Sham Comparator): Participants randomized to this group will follow a public Instagram account. This account was chosen because they have a strong following (over 600,000 followers) and it is a public account that anyone can follow. The content shared on this page is motivational and community driven. There is a focus of healthy living with an emphasis on exercise. Additionally, there are no paid sponsorships or radical exercise advice, which is common on other influencer pages. The Co-PIs determined that this page accurately represents the exercise-related content that is readily available on Instagram. The research team will not have control over the content of this account, but the account holder will be notified about the study.
  Interventions: Behavioral: Influencer Instagram account
- Student (Experimental): Student Co-PI will manage this Instagram account created for the study. Although the student is a Kinesiology student and works within the health field, she will not disclose this information on the account. Instead, she will present herself as a general college student. By withholding her major and career aspirations, we hope to get unbiased feedback on what participants think about the content being presented. The content presented will be identical to study arm #3.
  Interventions: Behavioral: Research study Instagram account
- Scientist (Experimental): The PI will manage this Instagram account created for the study. The PI is a certified exercise physiologist and holds a PhD in Rehabilitation Sciences. She will disclose this information on the account. This group is the study's "gold standard" because it will provide evidence-based content delivered by an exercise scientist.
  Interventions: Behavioral: Research study Instagram account

INTERVENTIONS:
Behavioral: Influencer Instagram account — Participants randomized to this group will follow a public Instagram account. This account was chosen because they have a strong following (over 600,000 followers) and it is a public account that anyone can follow. The content shared on this page is motivational and community driven. There is a focus of healthy living with an emphasis on exercise. Additionally, there are no paid sponsorships or radical exercise advice, which is common on other influencer pages. The Co-PIs determined that this page accurately represents the exercise-related content that is readily available on Instagram. The research team will not have control over the content of this account, but the account holder will be notified about the study.
  Arms: Control
Behavioral: Research study Instagram account — Intervention arms will deliver the same exercise-related content on the same schedule on the intervention Instagram accounts. The arms will deliver 13-weeks worth of content which goes through the last possible day of the intervention. The structure was based on feedback from stakeholders in a formative focus group. All of the content delivered through the accounts is evidence-based and referenced from reputation organizations/agencies such as the American College of Sports Medicine, American Heart Association, Center for Disease Control, and World Health Organization. Each Co-PI will post videos to answer participant questions. To ensure that the content between both groups is the same, the Co-PIs will meet to determine which questions to answer and draft the response.
  Arms: Scientist; Student

SUMMARY:
This study is a 3-arm randomized intervention to provide exercise education through Instagram. The primary outcome is trust in the content presented.

DETAILED DESCRIPTION:
Social media is an interpersonal-level technology that can provide physical activity support through social support and behavioral education. One popular social media platform is Instagram. However, there is limited data on whether participants trust the content delivered through this platform. There is also limited information on whether the social-media account holder plays a role in the acceptance of the content. The purpose of the proposed study is to determine participants perceptions of physical activity related information and social media account. The design for this study is a 3-arm randomized intervention through Instagram. Participants (n=60) will be randomized to one of three Instagram accounts (control, student, and scientist). Recruitment will be on a rolling basis for 2 months; once participants are deemed eligible, they will be enrolled for 4-weeks and will receive a weekly questionnaire to determine their perceptions. Participants will also be encouraged to participate in follow-up questionnaires at 2 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* less than 150 minutes of moderate-to-vigorous exercise per week
* active Instagram account

Exclusion Criteria:

* physical activity is inadvisable based on the PAR-Q+

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Self-reported trust in Instagram content assessed with a likert scale | 4-weeks
  Participant trust in the content presented on the Instagram account using a 10-point scale where 1 is low trust and 10 is high trust

SECONDARY OUTCOMES:
Physical activity measured by the IPAQ | 4-weeks
  self-reported total physical activity MET*minutes/week

CONTACTS AND LOCATIONS:
Locations (1):
- California State Polytechnic University, Pomona, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No